CLINICAL TRIAL: NCT03469674
Title: Randomised Phase III Trial of Molecular Profile-based Versus Standard Recommendations for Adjuvant Radiotherapy for Women With Early Stage Endometrial Cancer: PORTEC-4a Trial
Brief Title: PORTEC-4a: Molecular Profile-based Versus Standard Adjuvant Radiotherapy in Endometrial Cancer
Acronym: PORTEC-4a
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other); Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Principal Investigator, Carien Creutzberg, Chief Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P16.054; UL2011-5336 (Other Grant/Funding Number: Dutch Cancer Society); ISRCTN11659025 (Registry Identifier: ISRCTN Registry); NTR5841 (Registry Identifier: Netherlands Trials Registry)
Record Dates: First submitted 2018-03-08; First posted 2018-03-19 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Endometrial Cancer Stage I; Endometrial Cancer Stage II
Keywords: Radiotherapy; Vaginal brachytherapy; Molecular risk factors
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Observation

STUDY DESIGN:
Intervention Model Description: 2:1 randomisation to adjuvant treatment assignment based on the integrated molecular risk profile or standard adjuvant vaginal brachytherapy
Masking Description: Evaluation of outcomes is done without information on randomised arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molecular profile based treatment (Experimental): Determination of the integrated clinicopathological and molecular profile to determine adjuvant treatment: observation for favourable profile; vaginal brachytherapy for intermediate profile; external beam radiotherapy for unfavourable profile
  Interventions: Radiation: Vaginal brachytherapy; Radiation: External beam radiotherapy; Other: Observation
- Vaginal brachytherapy (Active Comparator): Adjuvant vaginal brachytherapy (standard treatment)
  Interventions: Radiation: Vaginal brachytherapy

INTERVENTIONS:
Radiation: Vaginal brachytherapy — Internal radiation of the vaginal vault using a vaginal cylinder, 21 Gy in 3 out-patient sessions over 2 weeks
Radiation: External beam radiotherapy — External beam pelvic radiotherapy on a linear accelerator, 48.6 Gy in 27 out-patients sessions over 5.5 weeks
  Arms: Molecular profile based treatment
Other: Observation — No radiation therapy, but active follow-up and quality of life questionnaires as in the groups who have adjuvant treatment
  Arms: Molecular profile based treatment

SUMMARY:
This is prospective, multicenter, randomised phase III trial among women with endometrial cancer with high-intermediate risk features to investigate the role of an integrated clinicopathological and molecular risk profile to determine if participants should receive no adjuvant therapy, vaginal brachytherapy or external beam radiotherapy based on a favourable, intermediate or unfavourable profile as compared to standard adjuvant vaginal brachytherapy.

DETAILED DESCRIPTION:
Adjuvant therapy for women with endometrial cancer has increasingly been tailored to prognostic factors to prevent overtreatment and select those women for adjuvant treatment who will have a clinically relevant reduction of the risk of relapse by the adjuvant treatment. Risk profiles have traditionally been based on clinicopathological factors such as age, stage, grade, LVSI and depth of invasion. Newer, both molecular-genetic (the cancer genome atlas subgroups) or immunohistochemistry-based (L1-CAM) risk factors have become available which are strongly related to outcomes and risk of cancer spread. In a comprehensive analysis of the PORTEC-1 and-2 biobank an integrated clinicopathological and molecular risk profile was determined which separated the current high-intermediate risk group of endometrial cancer in 3 separate groups (favourable, intermediate or unfavourable) with clearly separated outcomes, which is now prospectively tested in the clinic to determine adjuvant treatment. This is the first randomised trial using the molecular risk factors to assign adjuvant treatment for women with stage I-II high-intermediate risk endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrioid type endometrial carcinoma, International Federation of Gynecology and Obstetrics (FIGO) 2009 stage I, with one of the following combinations of stage, grade, age, and lymph-vascular space invasion (LVSI):

  1. Stage IA, grade 3 (any age, with or without LVSI)
  2. Stage IB, grade 1 or 2 and age >60 years
  3. Stage IB, grade 1-2 with documented LVSI
  4. Stage IB, grade 3 without LVSI
  5. Stage II (microscopic), grade 1
* World Health Organization (WHO)-performance status 0-2
* Written informed consent

Exclusion Criteria:

* Any other stage and type of endometrial carcinoma
* Histological types serous carcinoma or clear cell carcinoma (at least 10% if mixed type), or undifferentiated or neuroendocrine carcinoma
* Uterine sarcoma (including carcinosarcoma)
* Previous malignancy (except for non-melanomatous skin cancer) < 5 yrs
* Previous pelvic radiotherapy
* Expected interval between the operation and start of radiotherapy exceeding 8 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2016-06-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal recurrence | 5 years
  Total vaginal recurrence and vaginal recurrence as first failure

SECONDARY OUTCOMES:
Adverse events | 5 years
  Treatment-related symptoms according to CTCAE v 4.0
Health-related cancer-specific quality of life | 5 years
  Cancer-specific quality of life (European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (QLQC-30) - clinically relevant changes on QLQC30 functioning scales, general quality of life and general cancer symptoms
Endometrial cancer-related symptoms and quality of life | 5 years
  Endometrial cancer-related specific symptoms (EORTC EN24 module)- clinically relevant changes on these scales (quite a bit/very much vs no or mild symptoms)
Relapse-free survival | 5 years
  Relapse-free survival (survival without relapse)
Survival | 5 years
  Overall survival (all-cause death)
5-year vaginal control including treatment for relapse | 5 years
  Long-term local control including salvage treatment for local relapse
Pelvic recurrence (total) | 5 years
  Total pelvic recurrences
Pelvic recurrence as first failure | 5 years
  Pelvic recurrence as first failure
Distant recurrence (total) | 5 years
  Total distant recurrences
Distant recurrence as first failure | 5 years
  Distant recurrence as first failure
Endometrial cancer related health care costs | 5 years
  All hospital based health care costs used with primary treatment or during followup for treatment of adverse events and/or treatment for relapse

OTHER OUTCOMES:
Recurrence (vaginal and total) per risk profile | 5 years
  Vaginal, pelvic and distant relapse split by risk profile and compared between the 2 arms

CONTACTS AND LOCATIONS:
Overall Officials: Carien L. Creutzberg, MD, PhD, Study Chair — Leiden University Medical Center, Dept of Radiation Oncology; Remi A. Nout, MD, PhD, Principal Investigator — ErasmusMC Dept of Radiation Oncology; Anne-Sophie van den Heerik, MD, Principal Investigator — Leiden University Medical Center, Dept of Radiation Oncology
Locations (31):
- Medical University, Vienna, Vienna, Austria
- University Hospital Gent, Ghent, Belgium
- CEEGOG, General Faculty Hospital and First Faculty of Medicine, Charles University, Prague, Prague, Czechia
- France (3):
  - GINECO group - Institut Goustave Roussy, Paris
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital Tenon, Paris
- Germany (7):
  - Sankt Gertrauden Krankenhaus, Berlin
  - Kaiserswerther Diakonie, Düsseldorf
  - Evang. Kliniken Essen-Mitte, Essen
  - Universitatsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Rotkreuzklinikum München, Münich
  - University Hospital, Tübingen
- Ireland (2):
  - CancerTrials Ireland - St James Hospital (SLRON SJH), Dublin
  - CancerTrials Ireland - St Luke's Hospital (SLRON SLH), Dublin
- Netherlands (15):
  - Academic Medical Center, Amsterdam
  - NKI / Antoni van Leeuwenhoekhuis, Amsterdam
  - Radiation Therapy Group, Arnhem
  - Catharina Hospital, Eindhoven
  - Zuidwest Radiotherapy Institute, Flushing
  - University Medical Center Groningen, Groningen
  - Radiotherapy Institute Friesland, Leeuwarden
  - Leiden University Medical Center, Leiden
  - MAASTRO radiation oncology clinic, Maastricht
  - Radboud University Medical Center, Nijmegen
  - ErasmusMC Cancer Center, Rotterdam
  - Haaglanden Medical Center, The Hague
  - Verbeeten institute, Tilburg
  - University Medical Center Utrecht, Utrecht
  - Isala Clinics, Zwolle
- Kantonsspital Frauenklinik Lucerne, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Specifics will be decided and made public on website at a later stage, most probably from 5 years after final publication onwards
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From 5 years after final publication onwards
Access Criteria: Upon written application with a clear decription of aim, methods and analysis plan, publication plan, after approval from the study team

REFERENCES:
- [Derived] van den Heerik ASVM, Horeweg N, Haverkort MAD, Kuijsters N, Kommoss S, Koppe FLA, Nowee ME, Westerveld H, De Jong MAA, Fruhauf F, Cnossen JS, Mens JWM, Beukema JC, Chargari C, Gillham C, Jurgenliemk-Schulz IM, Vandecasteele K, Hamann M, Kiderlen M, Staebler A, Nijman HW, Wortman BG, Asteinidou E, de Boer SM, van den Hout WB, Verhoeven-Adema KW, Nout RA, Putter H, Bosse T, Creutzberg CL. Molecular profile-based adjuvant treatment for women with high-intermediate risk endometrial cancer (PORTEC-4a): results of a randomised, open-label, phase 3, multicentre, non-inferiority trial. Lancet Oncol. 2026 Jan;27(1):23-35. doi: 10.1016/S1470-2045(25)00612-6. PMID 41449145
- [Derived] Nero C, Ciccarone F, Pietragalla A, Duranti S, Daniele G, Scambia G, Lorusso D. Adjuvant Treatment Recommendations in Early-Stage Endometrial Cancer: What Changes With the Introduction of The Integrated Molecular-Based Risk Assessment. Front Oncol. 2021 Sep 1;11:612450. doi: 10.3389/fonc.2021.612450. eCollection 2021. PMID 34540651
- [Derived] van den Heerik ASVM, Horeweg N, Nout RA, Lutgens LCHW, van der Steen-Banasik EM, Westerveld GH, van den Berg HA, Slot A, Koppe FLA, Kommoss S, Mens JWM, Nowee ME, Bijmolt S, Cibula D, Stam TC, Jurgenliemk-Schulz IM, Snyers A, Hamann M, Zwanenburg AG, Coen VLMA, Vandecasteele K, Gillham C, Chargari C, Verhoeven-Adema KW, Putter H, van den Hout WB, Wortman BG, Nijman HW, Bosse T, Creutzberg CL. PORTEC-4a: international randomized trial of molecular profile-based adjuvant treatment for women with high-intermediate risk endometrial cancer. Int J Gynecol Cancer. 2020 Dec;30(12):2002-2007. doi: 10.1136/ijgc-2020-001929. Epub 2020 Oct 12. PMID 33046573
- [Derived] Wortman BG, Bosse T, Nout RA, Lutgens LCHW, van der Steen-Banasik EM, Westerveld H, van den Berg H, Slot A, De Winter KAJ, Verhoeven-Adema KW, Smit VTHBM, Creutzberg CL; PORTEC Study Group. Molecular-integrated risk profile to determine adjuvant radiotherapy in endometrial cancer: Evaluation of the pilot phase of the PORTEC-4a trial. Gynecol Oncol. 2018 Oct;151(1):69-75. doi: 10.1016/j.ygyno.2018.07.020. Epub 2018 Aug 3. PMID 30078506
- See also: Study website — http://www.msbi.nl/portec4